CLINICAL TRIAL: NCT04371653
Title: A Prospective, Randomized, Placebo-Controlled Pilot Study to Characterize the Intestinal Microbiome and to Evaluate the Safety and Fecal Microbiome Changes Following Twice Weekly Administration of Lyophilized PRIM-DJ2727 or Placebo Given Orally for 12 Weeks in Subjects With Nonalcoholic Fatty Liver Disease (NAFLD)
Brief Title: A Prospective, Randomized, Placebo-Controlled Pilot Study to Characterize the Intestinal Microbiome and to Evaluate the Safety and Fecal Microbiome Changes Following Administration of Lyophilized PRIM-DJ2727 or Placebo Given Orally in Subjects With Nonalcoholic Fatty Liver Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of funds
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Herbert DuPont, MD, Professor of Infectious Diseases, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-SPH-19-1126
Record Dates: First submitted 2020-04-22; First posted 2020-05-01 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Nonalcoholic Fatty Liver Disease (NAFLD) With History of Diabetes Melitus
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active group (Experimental): Patients with NAFLD will receive orally fecal microbiota capsules from healthy donors
  Interventions: Drug: PRIM-DJ2727
- Placebo group (Placebo Comparator): Placebo capsules will be identical to the active capsules, but not contain intestinal bacteria
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PRIM-DJ2727 — administration orally
  Arms: Active group
Drug: Placebo — administration orally placebo
  Arms: Placebo group

SUMMARY:
Potential subjects with non-alcoholic fatty liver disease (NAFLD) will be identified by gastroenterologists (study investigators). Twelve eligible subjects with NAFLD will be randomly assigned to receive either active fecal microbiota transplantation in orally administered capsules or Placebo capsules and dosed twice weekly for 12 weeks. .

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. For sexually active male and female subjects of childbearing potential, agree to use an effective method of birth control during the study.
3. For female subjects of childbearing potential, a negative urine Qualitative HCG pregnancy test at enrollment and on the Week 1, Day 1 of the Treatment prior to administration of study drug.
4. Willing and able to sign an informed consent form and attend study assessments and follow up visits.
5. A documented diagnosis of NAFLD without cirrhosis based on imaging or clinical judgment of a gastroenterologist or hepatologist.
6. History of diabetes mellitus
7. Has an attending physician who will provide non-transplant care for the subject.
8. Agrees to maintain a stable regimen including weight loss, exercise, medications to control lipids and glucose, and vitamin E therapy if already prescribed, during participation in the study

Exclusion Criteria:

1. Unable to take multiple capsules orally.
2. Alcohol consumption of greater than an average of one drink per day for women and two drinks per day for men.
3. Hemochromatosis.
4. Hepatic encephalopathy.
5. Compromised immune system (e.g. primary immune disorders or clinical immunosuppression due to a medical condition or medication e.g. taking oral prednisone >20 mg a day or prednisone-equivalent)
6. Receipt of systemic non-topical antibiotic therapy within 14 days of treatment day 1.
7. History of use of an investigational drug within 90 days prior to the screening visit.
8. Positive results for active HIV, Hepatitis B, or Hepatitis C infections.
9. Current history for active states of Inflammatory bowel disease, Irritable bowel syndrome, microscopic colitis, celiac disease, short gut syndrome, colostomy, colectomy, gastrointestinal fistulae or strictures.
10. History of significant uncontrolled systemic disease that in the opinion of the study investigator could interfere with study participation and/or objectives.
11. Life expectancy of < 1 year.
12. In the opinion of investigator, subject for any reason, should be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Microbiome Diversity in Fecal Samples as Indicated by the Shannon Diversity Index | 10 months
  The Shannon diversity index is used to characterize species diversity in a community. Shannon's index accounts for both abundance and evenness of the species present. A high index value would represent a diverse and equally distributed community, and lower values represent a less diverse community. A value of 0 would represent a community with just one species. Typical values are generally between 1.5 and 3.5.
Microbiome Richness in Fecal Samples as Indicated by the Number of Taxonomies per Participant | 10 months
Number of Participants With an Increase in Flora Diversity in Fecal Samples | 10 months

SECONDARY OUTCOMES:
Changes in gut motility | 6 months
  Changes in gut motility will be determined using Smart Pill (if completed successfully pre and post treatment) measuring gut motility
Monitor subjects' health information | 10 months
  The SF-36 will be administered at enrollment, follow-up clinic visits at Week 13 and 9 month, and early termination visit. Rapid Eating Assessment for Patients (REAP) is to help quickly assess diet and physical activity of individuals. In addition, subjects will be asked to maintain a paper diary recording number of BM per day and type of each BM after enrollment. Information such as hospitalizations or mortality from any cause will be collected as part of the health outcomes assessment throughout this study.

IPD SHARING:
Plan to Share IPD: Undecided